CLINICAL TRIAL: NCT02826811
Title: Role of Anti-BK Virus Neutralizing Antibodies (BKV) as a Prognostic Marker for the Development of Nephropathy BK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6368
Record Dates: First submitted 2016-06-15; First posted 2016-07-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-04

CONDITIONS: Graft Dysfunction
Keywords: Graft dysfunction; Graft loss; kidney; Transplantation; BKV; Anti-BKV; Nephropathy; Immunosuppression; Prognostic markers
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
BKV nephropathy (BKV) is one of the most frequent complications of kidney transplantation.

In the absence of specific anti-BKV treatment, pre-emptive reduction of immunosuppression is the main strategy that has proven effective in reducing the risk of BKVN. However, it exposes a transplant rejection risk estimated between 4 and 14% according to studies.

Despite the pre-emptive reduction of immunosuppression, a significant number of patients continue to progress towards BKVN suggesting that pre-emptive strategy is late. It's therefore urgent to develop new prognostic markers to identify earlier and more effectively patients with a higher risk of developing BKVN.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Grafted kidney patient between 1 July 2012 and 31 July 2014 at Strasbourg University Hospital with regular monitoring

Exclusion Criteria:

* Patient under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients between 1 July 2012 and 31 July 2014 at the University Hospital of Strasbourg
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Quantification of anti-BKV | up to 12 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Samira FAFI-KREMER, PharmD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Virologie - Hôpital Civil, Strasbourg, France, France

IPD SHARING:
Plan to Share IPD: No